CLINICAL TRIAL: NCT04185129
Title: Comparison Efficacy in Patients With Asthma Using Foster MDI and Relvar Medications
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Far Eastern Memorial Hospital (Other)
Collaborators: Orient Europharma Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Shih-Lung Cheng, MD. PhD, Far Eastern Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Foster 001
Record Dates: First submitted 2019-11-28; First posted 2019-12-04 (Actual); Last update posted 2019-12-04 (Actual); Status verified 2019-12

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Foster Home Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Foster (Experimental): uncontrolled asthma patients were randomized into Foster treatment group
  Interventions: Drug: Foster
- Relvar (Active Comparator): uncontrolled asthma patients were randomized into Relvar treatment group
  Interventions: Drug: Foster

INTERVENTIONS:
Drug: Foster — a randomized study for comparison asthma patients using Foster or Relvar. The primary end point is lung function improvement evaluation
  Other Names: Relvar

SUMMARY:
This is a randomized study to compare asthma patients using Foster or Relvar.

DETAILED DESCRIPTION:
The Global Asthma Association (GAA) and the World Allergy Organization (WAO) recently issued statements stating that the small airway is caused by asthma and chronic obstructive pulmonary disease (COPD). Both pathogenesis and treatment play an important role. The small airway is an airway with diameter less than 2 mm and is one of the main sites where airflow obstruction occurs. Small particles (<2 μm) and large particles are more likely to deposit in the distal airways, and have shown to have better effects on asthma and pulmonary obstruction. At the same time, real-life research has also shown that extra-fine particles provide better asthma control than large particles, and can better improve quality of life.The aim of the study is to compare the efficacy of asthma inhalers between extra-fine particles and non-extra-fine particles.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosis with asthma with treatment naive
* asthma patients with poor controlled status

Exclusion Criteria:

* COPD
* smoking history
* pregnancy
* cardiaovascular disease
* patients with acute respiratory infection

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Lung function improvement | one year
  FEV1

CONTACTS AND LOCATIONS:
Overall Officials: Shih-Lung Cheng, Principal Investigator — Far Eastern Memorial Hospital
Locations (1):
- Far Eastern Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No